CLINICAL TRIAL: NCT00824564
Title: Prospective Randomized Phase IV Open Label Comparative Study Of Tranexamic Acid Plus Standard Of Care Versus Standard Of Care For The Reduction Of Blood Loss In Patients Undergoing Surgery For Long Bone Fracture
Brief Title: Study Of Tranexamic Acid For The Reduction Of Blood Loss In Patients Undergoing Surgery For Long Bone Fracture
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B1461002
Record Dates: First submitted 2009-01-14; First posted 2009-01-16 (Estimated); Results first posted 2011-06-28 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Femoral Fractures
Keywords: Tranexamic Acid; Blood Loss; Long Bone Fracture Surgery
MeSH Terms: conditions — Femoral Fractures; Hemorrhage | interventions — Tranexamic Acid; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Tranexamic Acid plus standard of care
  Interventions: Drug: Tranexamic Acid plus standard of care
- B (Other): Standard of care includes the routine surgical and anesthetic techniques being utilized to control blood loss.
  Interventions: Procedure: Standard of care

INTERVENTIONS:
Drug: Tranexamic Acid plus standard of care — Tranexamic acid given slowly intravenously (15 mg/kg body weight) 15 minutes before surgery followed by a second dose at three hour interval from first dose and third dose at three hour interval from the second + Standard of care (Standard of care includes the routine surgical and anesthetic techniques being utilized to control blood loss)
  Arms: A
Procedure: Standard of care — Standard of care includes the routine surgical and anesthetic techniques being utilized to control blood loss
  Arms: B

SUMMARY:
Tranexamic acid has been shown to reduce postoperative blood losses and transfusion requirements in a number of types of surgery. Most trials in orthopedic surgery have been conducted in arthroplasty, hip fracture and spine surgeries. This study would aim to see the effect of tranexamic acid in reduction of blood loss and transfusions for long bone fracture surgery, primarily fracture shaft of femur.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing surgery for fracture shaft of femur

Exclusion Criteria:

* Patients with a platelet count less than 100, 000/mm3 or history of thrombocytopenia
* Patients with known coagulopathy
* Patients with anemia (hemoglobin levels less than 8 mg/dl or hematocrit <24%)
* Patients with documented DVT or PE at screening or in past three months
* Patients having known hypersensitivity to tranexamic acid or any other constituent of the product
* Patients with any associated major illness (e.g., severe cardiac or respiratory disease)
* Anticoagulants (other than LMWH or heparin in prophylactic doses to prevent deep vein thrombosis), direct thrombin inhibitors or thrombolytic therapy administered or completed within last week

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2009-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Coimbatore, Tamil Nadu, India

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1461002&StudyName=Study%20Of%20Tranexamic%20Acid%20For%20The%20Reduction%20Of%20Blood%20Loss%20In%20Patients%20Undergoing%20Surgery%20For%20Long%20Bone%20Fracture

RESULTS

PARTICIPANT FLOW:
Groups:
- Tranexamic Acid Plus Standard of Care: Tranexamic acid given slowly intravenously (IV) (15 milligram (mg) / kilogram (kg) body weight) 15 minutes before surgery followed by a second dose at 3 hour interval from first dose and third dose at 3 hour interval from the second + Standard of care (included the routine surgical and anesthetic techniques being utilized to control blood loss).
- Standard of Care: Standard of care included the routine surgical and anesthetic techniques being utilized to control blood loss.
Period: Overall Study
Arm/Group | Tranexamic Acid Plus Standard of Care | Standard of Care
Started | 42 | 40
Treated | 41 | 40
Completed | 34 | 30
Not Completed | 8 | 10
Not completed — Lost to Follow-up | 5 | 7
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Other | 1 | 2
Not completed — Randomized, but not treated | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tranexamic Acid Plus Standard of Care | Standard of Care | Total
Number analyzed (Participants) | 41 | 40 | 81
Age Continuous [Mean (Standard Deviation); unit: Years] | 33.7 (12.6) | 36.6 (17.0) | 35.1 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 36 | 33 | 69

OUTCOME MEASURES:

1. Primary Outcome: Total Blood Loss
Description: Total blood loss was defined as the sum of intra-operative and post-operative blood loss. It was measured by weighing the drapes/ dressings or swabs prior to soaking to measure difference in weight and checking drain collectors until drains were removed.
Time Frame: Baseline through Day 7 post-surgery
Population: Full analysis set (FAS) included all participants who were randomized to study treatment and received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: Milliliters (mL)
Arm/Group | Tranexamic Acid Plus Standard of Care | Standard of Care
Number analyzed (Participants) | 41 | 40
Milliliters (mL) | 370.7 (180.7) | 426.2 (323.8)
Statistical Analysis 1: Comparison: Tranexamic Acid Plus Standard of Care vs Standard of Care; The mean difference with associated standard error (SE), and corresponding 95% confidence interval (CI) for the comparisons of tranexamic acid plus standard of care against Standard of care was presented along with the p-value for the test. Two-sample t-test was performed at 5% level of significance; Test type: Superiority or Other; p = 0.348, t-test, 2 sided; Mean Difference (Final Values) = -55.5, 95% CI 2-sided [-172.7 to 61.7], Standard Error of Mean 58.63

2. Secondary Outcome: Intra-operative Blood Loss
Description: Intra-operative blood loss was measured by weighing the drapes/ dressings or swabs prior to soaking to measure difference in weight and checking drain collectors until drains were removed.
Time Frame: Day 1 (End of surgery)
Population: FAS included all participants who were randomized to study treatment and received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Tranexamic Acid Plus Standard of Care | Standard of Care
Number analyzed (Participants) | 41 | 40
mL | 316.2 (129.8) | 292.2 (161.6)
Statistical Analysis 1: Comparison: Tranexamic Acid Plus Standard of Care vs Standard of Care; The mean difference with associated SE and corresponding 95% CI for the comparisons of tranexamic acid plus standard of care against Standard of care was presented along with the p-value for the test. Two-sample t-test was performed at 5% level of significance; Test type: Superiority or Other; p = 0.466, t-test, 2 sided; Mean Difference (Final Values) = 24.0, 95% CI 2-sided [-41.3 to 89.3], Standard Error of Mean 32.78

3. Secondary Outcome: Post-operative Blood Loss
Description: Post-operative blood loss was defined as the sum of the drainage volumes measured over post-operative days 1, 2, and at drain removal. It was measured by weighing the drapes/ dressings or swabs prior to soaking to measure difference in weight and checking drain collectors until drains were removed.
Time Frame: 1, 4, 8 and 24 hours post-surgery
Population: FAS included all participants who were randomized to study treatment and received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Tranexamic Acid Plus Standard of Care | Standard of Care
Number analyzed (Participants) | 41 | 40
mL
  1 hour | 0.2 (1.6) | 9.5 (35.6)
  4 hours | 0.6 (3.2) | 7.4 (20.5)
  8 hours | 0.7 (3.5) | 7.5 (26.7)
  24 hours | 27.4 (67.5) | 50.1 (68.9)
Statistical Analysis 1: Comparison: Tranexamic Acid Plus Standard of Care vs Standard of Care; For 1 hour post-surgery, the mean difference with associated SE and corresponding 95% CI for the comparisons of tranexamic acid plus standard of care against Standard of care was presented along with the p-value for the test. Two-sample t-test was performed at 5% level of significance; Test type: Superiority or Other; p = 0.109, t-test, 2 sided; Mean Difference (Final Values) = -9.3, 95% CI 2-sided [-20.7 to 2.2], Standard Error of Mean 5.57
Statistical Analysis 2: Comparison: Tranexamic Acid Plus Standard of Care vs Standard of Care; For 4 hour post-surgery, the mean difference with associated SE, and corresponding 95% CI for the comparisons of tranexamic acid plus standard of care against Standard of care was presented along with the p-value for the test. Two-sample t-test was performed at 5% level of significance; Test type: Superiority or Other; p = 0.045, t-test, 2 sided; Mean Difference (Final Values) = -6.8, 95% CI 2-sided [-13.4 to -0.1], Standard Error of Mean 3.24
Statistical Analysis 3: Comparison: Tranexamic Acid Plus Standard of Care vs Standard of Care; For 8 hour post-surgery, the mean difference with associated SE, and corresponding 95% CI for the comparisons of tranexamic acid plus standard of care against Standard of care was presented along with the p-value for the test. Two-sample t-test was performed at 5% level of significance; Test type: Superiority or Other; p = 0.119, t-test, 2 sided; Mean Difference (Final Values) = -6.8, 95% CI 2-sided [-15.4 to 1.8], Standard Error of Mean 4.20
Statistical Analysis 4: Comparison: Tranexamic Acid Plus Standard of Care vs Standard of Care; For 24 hour post-surgery, the mean difference with associated SE, and corresponding 95% CI for the comparisons of tranexamic acid plus standard of care against Standard of care was presented along with the p-value for the test. Two-sample t-test was performed at 5% level of significance; Test type: Superiority or Other; p = 0.139, t-test, 2 sided; Mean Difference (Final Values) = -22.7, 95% CI 2-sided [-52.9 to 7.5], Standard Error of Mean 15.16

4. Secondary Outcome: Total Blood Loss Assessed by Gross' Formula
Description: Gross's formula for estimating total blood loss: Estimated blood volume*[(Hematocrit initial - Hematocrit final)/ Hematocrit average]; where estimated blood volume equals body weight in kilograms (kg) *70 mL/kg.
Time Frame: Day 7 post-surgery
Population: FAS included all participants who were randomized to study treatment and received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Tranexamic Acid Plus Standard of Care | Standard of Care
Number analyzed (Participants) | 41 | 40
mL | 823.2 (676.6) | 798.0 (490.2)
Statistical Analysis 1: Comparison: Tranexamic Acid Plus Standard of Care vs Standard of Care; The mean difference with associated SE, and corresponding 95% CI for the comparisons of tranexamic acid plus standard of care against Standard of care was presented along with the p-value for the test. Two-sample t-test was performed at 5% level of significance; Test type: Superiority or Other; p = 0.849, t-test, 2 sided; Mean Difference (Final Values) = 25.2, 95% CI 2-sided [-238.2 to 288.6], Standard Error of Mean 132.10

5. Secondary Outcome: Number of Participants Receiving Transfusions
Description: A uniform transfusion protocol was maintained for all participants in the study. Transfusion to be triggered at 8.0 milligram/deciliter (mg/dl) hemoglobin or haematocrit value of 24 percent.
Time Frame: Up to day 7 post-surgery
Population: FAS included all participants who were randomized to study treatment and received at least one dose of study medication.
Measure: Number (95% Confidence Interval); unit: Participants
Arm/Group | Tranexamic Acid Plus Standard of Care | Standard of Care
Number analyzed (Participants) | 41 | 40
Participants | 5 [4.1 to 26.2] | 6 [5.7 to 29.8]
Statistical Analysis 1: Comparison: Tranexamic Acid Plus Standard of Care vs Standard of Care; Chi-square test was used at 5% level of significance; Test type: Superiority or Other; p = 0.714, Chi-squared

6. Secondary Outcome: Change From Baseline in Hemoglobin Levels at End of Surgery, 1 hr Post-surgery, and Mornings of Day 1, Day 2, Day 4, Day 7 or Early Termination (ET) Post-surgery
Time Frame: Baseline through end of surgery, 1 hr post-surgery, and mornings of Day 1, Day 2, Day 4, Day 7 or ET post-surgery
Population: FAS included all participants who were randomized to study treatment and received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: gram/deciliter (g/dl)
Arm/Group | Tranexamic Acid Plus Standard of Care | Standard of Care
Number analyzed (Participants) | 41 | 40
gram/deciliter (g/dl)
  Baseline | 13.1 (1.5) | 12.9 (2.1)
  Change at end of surgery | -1.7 (1.2) | -2.0 (1.5)
  Change at 1 hour post-surgery | -1.8 (1.1) | -1.9 (1.3)
  Change at day 1 post-surgery | -2.1 (1.1) | -2.2 (1.4)
  Change at day 2 post-surgery | -2.1 (1.2) | -2.3 (1.4)
  Change at day 4 post-surgery or ET | -2.0 (1.4) | -2.1 (1.5)
Statistical Analysis 1: Comparison: Tranexamic Acid Plus Standard of Care vs Standard of Care; For change at end of surgery, a Mixed Model Repeated Measures (MMRM) approach was used to relate the dependent (outcome) variable and independent (treatment, time point, and treatment-by-time point interaction as factors and baseline value as co-variate) variables taking into account the within-participant correlation arising from the repeated measurements; Test type: Superiority or Other; p = 0.208, Mixed Models Analysis; Least square means difference = 0.37, 95% CI 2-sided [-0.21 to 0.96], Standard Error of Mean 0.295
Statistical Analysis 2: Comparison: Tranexamic Acid Plus Standard of Care vs Standard of Care; For change at 1 hour post-surgery, a MMRM approach was used to relate the dependent (outcome) variable and independent (treatment, time point, and treatment-by-time point interaction as factors and baseline value as co-variate) variables taking into account the within-participant correlation arising from the repeated measurements; Test type: Superiority or Other; p = 0.682, Mixed Models Analysis; Least square means difference = 0.10, 95% CI 2-sided [-0.40 to 0.61], Standard Error of Mean 0.255
Statistical Analysis 3: Comparison: Tranexamic Acid Plus Standard of Care vs Standard of Care; For change at day 1 post-surgery, a MMRM approach was used to relate the dependent (outcome) variable and independent (treatment, time point, and treatment-by-time point interaction as factors and baseline value as co-variate) variables taking into account the within-participant correlation arising from the repeated measurements; Test type: Superiority or Other; p = 0.569, Mixed Models Analysis; Least square means difference = 0.14, 95% CI 2-sided [-0.35 to 0.63], Standard Error of Mean 0.244
Statistical Analysis 4: Comparison: Tranexamic Acid Plus Standard of Care vs Standard of Care; For change at day 2 post-surgery, a MMRM approach was used to relate the dependent (outcome) variable and independent (treatment, time point, and treatment-by-time point interaction as factors and baseline value as co-variate) variables taking into account the within-participant correlation arising from the repeated measurements; Test type: Superiority or Other; p = 0.413, Mixed Models Analysis; Least square means difference = 0.20, 95% CI 2-sided [-0.29 to 0.70], Standard Error of Mean 0.249
Statistical Analysis 5: Comparison: Tranexamic Acid Plus Standard of Care vs Standard of Care; For change at day 4/ET post-surgery, a MMRM approach was used to relate the dependent (outcome) variable and independent (treatment, time point, and treatment-by-time point interaction as factors and baseline value as co-variate) variables taking into account the within-participant correlation arising from the repeated measurements; Test type: Superiority or Other; p = 0.686, Mixed Models Analysis; Least square means difference = 0.11, 95% CI 2-sided [-0.44 to 0.66], Standard Error of Mean 0.276

7. Secondary Outcome: Number of Participants With Deep Vein Thrombosis (DVT) Post Surgery
Description: DVT was defined if a segment of the deep vein of the lower limb was not compressible or a previous compressive vein became non compressive or there was no flow in the underlying vessel. Symptoms of DVT included pain in the lower limb, localized tenderness, swelling and warmth.
Time Frame: Day 5 post-surgery
Population: FAS included all participants who were randomized to study treatment and received at least one dose of study medication.
Measure: Number (95% Confidence Interval); unit: Participants
Arm/Group | Tranexamic Acid Plus Standard of Care | Standard of Care
Number analyzed (Participants) | 41 | 40
Participants | 3 [1.5 to 19.9] | 0 [0.0 to 8.8]
Statistical Analysis 1: Comparison: Tranexamic Acid Plus Standard of Care vs Standard of Care; Fisher's exact test at 5% level of significance was used as the event rate was low and the expected count for any cell in the (unstratified) 2*2 contingency table was less than 5; Test type: Superiority or Other; p = 0.241, Fisher Exact

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Tranexamic Acid Plus Standard of Care | Standard of Care
Serious Adverse Events (participants affected / at risk) | 4/41 | 1/40
Other Adverse Events (participants affected / at risk) | 28/41 | 26/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tranexamic Acid Plus Standard of Care (N=41) | Standard of Care (N=40)
Cardiac failure (Cardiac disorders) | 0 | 1
Fat embolism (Injury, poisoning and procedural complications) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tranexamic Acid Plus Standard of Care (N=41) | Standard of Care (N=40)
Vision blurred (Eye disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 7
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 5 | 1
Chest pain (General disorders) | 0 | 1
Chills (General disorders) | 1 | 2
Oedema peripheral (General disorders) | 0 | 2
Pain (General disorders) | 17 | 17
Pyrexia (General disorders) | 3 | 3
Excoriation (Injury, poisoning and procedural complications) | 0 | 1
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 5
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 3 | 2
Dysuria (Renal and urinary disorders) | 2 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 3 | 5
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The data for hemoglobin levels was planned but not evaluated on the morning of Day 7 post-surgery.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.